CLINICAL TRIAL: NCT02940795
Title: Maternal Transmission of Dietary Sugars in Breast Milk
Brief Title: Dietary Sugars Found In Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, David A. Fields, PhD, Associate Professor, University of Oklahoma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 5297
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Lactation
Keywords: breast feeding; fructose
MeSH Terms: conditions — Breast Feeding | interventions — Coke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coke cola (Experimental): Exclusively lactating mothers with infants between 4-6 weeks were investigated. Lactating mothers will be consume a 20 ounce bottle of coke cola.
  Interventions: Other: Coke; Other: Diet Rite
- Diet Rite (Experimental): Exclusively lactating mothers with infants between 4-6 weeks were asked to consume a 12 ounce bottle of diet rite.
  Interventions: Other: Coke; Other: Diet Rite

INTERVENTIONS:
Other: Coke — Patients were given a 20 ounce bottle of Coke Cola.
Other: Diet Rite — Patients were given a 12 ounce can of Diet Rite.

SUMMARY:
The majority of pregnant women in the United States are either overweight or obese at conception with their offspring having greater adiposity at birth, a 2-fold greater risk of later obesity and neonatal insulin resistance.

Conventional wisdom holds that breast-milk composition is uniform; recently our group has questioned this. An increase in consumption of dietary sugars including fructose over the past 30 years has risen, and this has been associated with chronic metabolic and endocrine disorders and phenotypic alterations that promote obesity and diabetes. However, no prior studies have examined how maternal increases of sugars/fructose during lactation affects breast-milk composition with potential transmission to the infant. The objective of this proposal is to comprehensively assess the presence and pharmacokinetics of sugars, including fructose in human breast-milk in response to maternal consumption. The central hypothesis is that a graded, dose-response relationship be-tween maternal adiposity and sugar concentrations in breast-milk exist and that milk fructose concentrations are associated with altered body composition in the first months of life. This proposal, guided by compelling preliminary data will examine the evidence linking high intakes of milk fructose with altered metabolism and early obesity by pursuing two Specific Aims: 1) Test novel relationships between breast-milk sugars and changes in infant fat mass and 2) Characterize the pharmacokinetics of milk sugars after consuming a 20 oz. cola. These aims are significant given the intractability of obesity/diabetes and a potentially identifiable novel target, making for a clear but powerful public message to reduce sugary beverage consumption during lactation.

DETAILED DESCRIPTION:
One of the most highly effective preventive measures a mother can make in protecting the health of her infant and herself is to breastfeed. Despite extensive research on breast-milk, limited information beyond basic micro/macronutrient composition currently exists in the literature. Breast-milk is a complex, non-uniform biological substance. In prior studies the PI has shown significant associations be-tween non-nutritive constituents in breast-milk (e.g. IL-6, TNF-α, insulin, leptin) and body composition in infants starting at 4wks of age. The putative causal influence of breastfeeding reducing obesity is mixed with no clear probative evidence showing causal pathways. Despite many studies in this area, there are no detailed studies that have examined the potential modifying role of maternal diet, especially one high in sugars on the compositional makeup of the three largest breast-milk sugars (glucose, galactose and lactose) with none to date looking at fructose. Animal models have demonstrated that the obesogenic effect of maternal fructose consumption is transmitted to offspring via breast-milk with fructose-fed lactating dams producing offspring with double fasting insulin levels compared to control pups. This is relevant in humans because of the increase in dietary sugar consumption that has occurred in the population.

A mother/infant cohort (n=37) has been established with detailed infant phenotypic body composition (dual-energy X-ray absorptiometry) and detailed breast-milk analysis (insulin, leptin, IL-6, TNF-α but no milk sugars other than glucose) in exclusively breast feeding mothers varying widely in BMI (19 to 44 kg/m2). Sampling of breast-milk and infant body composition occurred at both 4 and 24wks. As a proof of concept, fructose was detected in breast-milk from 9 of these mothers which was significantly related to infant body fat, which is a novel finding to date and has never been reported in the literature. Building upon this prior work this study will determine the concentration and pharmacokinetics of breast-milk sugars after a test beverage is consumed.

ELIGIBILITY:
Inclusion Criteria:

* Exclusively lactating mothers
* Mothers must be 3 weeks to 6 weeks postpartum

Exclusion Criteria:

* Smoked during pregnancy or are currently smoking
* Unable to provide breast milk samples using a breast pump

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fructose in breast milk will be measured in human breast milk at one month. | One month
  Breast milk fructose at one month will be analyzed.
The change in fructose in breast milk from one to six months. | Six months
  The potential change in breast milk fructose from one to six months will be investigated.

SECONDARY OUTCOMES:
Breast milk fructose will be measured after the ingestion of a regular 20 ounce bottle of coke and a 12 ounce can of diet rite. | 6 hours.
  After the ingestion of either a regular 20 ounce bottle of coke or a 12 ounce can of diet rite at ~ 6:00 am a milk sample will be obtained every hour until 12:00 pm.

CONTACTS AND LOCATIONS:
Overall Officials: David A Fields, PhD, Principal Investigator — University of Oklahoma

IPD SHARING:
Plan to Share IPD: No
No there is not a plan to share data.

REFERENCES:
- [Derived] Rother KI, Sylvetsky AC, Walter PJ, Garraffo HM, Fields DA. Pharmacokinetics of Sucralose and Acesulfame-Potassium in Breast Milk Following Ingestion of Diet Soda. J Pediatr Gastroenterol Nutr. 2018 Mar;66(3):466-470. doi: 10.1097/MPG.0000000000001817. PMID 29077645